CLINICAL TRIAL: NCT03165422
Title: A Real-World Study of Ipilimumab Treatment After Nivolumab Treatment in Melanoma in Japan
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-9DA
Record Dates: First submitted 2017-05-16; First posted 2017-05-24 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adult patients with melanoma: Adult patients with melanoma at participating centers in Japan
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional

SUMMARY:
This is a medical chart review of ipilimumab treatment after nivolumab treatment in melanoma in Japan

ELIGIBILITY:
Inclusion Criteria:

* Adult patients > 18 years of age or older
* Diagnosis of advanced melanoma (unresectable/metastatic), alive or deceased as of date of data collection
* Treated with ipilimumab between 31-Aug-2015 and 31-Mar-2017 before or after nivolumab treatment

Exclusion Criteria:

* Patients enrolled in any clinical trials at any time
* Overlapping use of nivolumab and ipilimumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with melanoma who are patients at the participating centers in Japan will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-12-29 (Actual); Study Completion 2018-12-29 (Actual)

PRIMARY OUTCOMES:
Incidence of ipilimumab treatment after nivolumab treatment | Approximately 19 months
Incidence of nivolumab treatment after ipilimumab treatment | Approximately 19 months
Duration of nivolumab treatment | Approximately 19 months
Duration of ipilimumab treatment | Approximately 19 months
Duration of interval between nivolumab treatment and ipilimumab treatment | Approximately 19 months

SECONDARY OUTCOMES:
overall response rate (ORR) | Approximately 19 months
best overall response rate (BORR) | Approximately 19 months
overall survival (OS) | Approximately 19 months
progression-free survival (PFS) | Approximately 19 months
incidence of treatment-related adverse events (AEs) | Approximately 19 months
  incidence of treatment-related adverse events (AEs)/adverse reactions (ARs)
severity of treatment-related adverse events (AEs) | Approximately 19 months
  severity of treatment-related adverse events (AEs)/adverse reactions (ARs)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Minato-ku, Tokyo, Japan

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm